CLINICAL TRIAL: NCT00904735
Title: IMATINIB Plus Hydroxyurea in the Treatment of Recurrent or Progressive Meningiomas: a Randomized Phase II Study
Brief Title: Hydroxyurea With or Without Imatinib Mesylate in Treating Patients With Recurrent or Progressive Meningioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Scientifico H. San Raffaele (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: SRSI-GICNO-08-002; CDR0000641101 (Registry Identifier: PDQ (Physician Data Query)); NOVARTIS-SRSI-GICNO-08-002
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult grade I meningioma; adult grade II meningioma; adult anaplastic meningioma; adult papillary meningioma; recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Meningioma; Brain Neoplasms | interventions — Hydroxyurea; Imatinib Mesylate

ARMS (2):
- Arm I (Experimental): Patients receive oral hydroxyurea twice daily and oral imatinib mesylate once daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: hydroxyurea; Drug: imatinib mesylate
- Arm II (Experimental): Patients receive oral hydroxyurea twice daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: hydroxyurea

INTERVENTIONS:
Drug: hydroxyurea — Given orally
Drug: imatinib mesylate — Given orally
  Arms: Arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as hydroxyurea, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether hydroxyurea is more effective when given alone or together with imatinib mesylate in treating patients with meningioma.

PURPOSE: This randomized phase II trial is studying how well hydroxyurea works compared with giving hydroxyurea together with imatinib mesylate in treating patients with recurrent or progressive meningioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the progression-free survival of patients with recurrent or progressive meningiomas treated with hydroxyurea with vs without imatinib mesylate after surgery and radiotherapy.

Secondary

* Determine the overall survival, and response rate of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to WHO grade (I vs II-III). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral hydroxyurea twice daily and oral imatinib mesylate once daily in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral hydroxyurea twice daily in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with meningioma

  * WHO grade I-III
* Recurrent or progressive disease after prior surgery and radiotherapy, or radiosurgery
* Not amenable to further surgery
* No optic nerve sheet tumor and neurofibromatosis type II
* No known brain metastasis

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* ANC > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin ≥ 9 mg/dL (transfusion allowed)
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* SGOT and SGPT < 2.5 times ULN
* Creatinine < 1.5 times ULN
* Negative pregnancy test
* Fertile patients must use effective barrier method contraception during and for up to 3 months after completion of study therapy
* No second malignancy
* No known chronic liver disease (i.e., active hepatitis, cirrhosis)
* No known HIV infection
* No significant history of non-compliance to medical regimens or inability to grant reliable informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent enzyme-inducing anti-epileptic drugs
* No concurrent therapeutic anticoagulation with warfarin (e.g., Coumadin®)

  * Low-molecular weight heparin (e.g., Lovenox) or heparin allowed
  * Mini-dose Coumadin® (e.g., 1 mg QD) allowed for prophylaxis of central venous catheter thrombosis, at the discretion of the treating physician
* No concurrent acetaminophen (Efferalgan®, Tachipirina®) allowed during imatinib mesylate administration
* No other concurrent anticancer agents, including chemotherapy or biological agents
* No other concurrent investigational drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2009-06

PRIMARY OUTCOMES:
Progression-free survival, defined as ≥ 25% increase in tumor volume or new tumor on MRI

SECONDARY OUTCOMES:
Survival
Response rate according to MacDonald criteria
Toxicity as assessed by NCI CTCAE v. 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Alba A. Brandes, MD, Study Chair — Ospedale Bellaria
Locations (5):
- Italy (5):
  - Ospedale Civile Avellino, Avellino
  - Ospedale Bellaria, Bologna
  - Azienda Ospedaliero Careggi, Florence
  - Istituto Nazionale Neurologico Carlo Besta, Milan
  - Ospedale Civile di Rovigo, Rovigo